CLINICAL TRIAL: NCT07205653
Title: Validity of Patients' Self-assessment of Tonsil Size
Brief Title: Self-assessment of Tonsil Size
Status: Not yet recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Henrik Sjöblom, Dr, Turku University Hospital
Other Study IDs: T2025/10790
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Tonsillar Hypertrophy
Keywords: tonsil size; tonsillar hypertrophy; self-assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The participants receive instructions on two tonsil size classification scales and then, using a tongue depressor as well as their mobile phone camera and/or a flashlight and a mirror, the participants assess the size of their own tonsils on two scales.

After the self-assessment, a medical student and two ear, nose, and throat (ENT) specialists evaluate the participants' tonsil size using a tongue depressor and a headlamp, applying the same scales.

The objective of this study is to demonstrate that patient self-assessment constitutes a sufficiently accurate method for evaluating tonsil size. Furthermore, it aims to show that patients experiencing conditions such as sleep apnea or swallowing difficulties can, on the basis of their own assessment, be appropriately referred to an otolaryngologist for surgical evaluation, thereby conserving healthcare resources and reducing the time burden for patients.

DETAILED DESCRIPTION:
A total of 70 to 100 medical students from the first to third year of study will be recruited beginning in 2025, with recruitment extended into 2026 if necessary. Participants will be provided with a plain-language summary of the research plan and will be asked to provide written informed consent to participate.

The investigators hypothesize that both participants and a trained medical student will be able to assess tonsil size-categorizing them as small, medium, or large, as well as grading them on a 0-4 scale-with sufficient agreement compared to professional evaluation, defined as an intraclass correlation coefficient (ICC) of at least 0.60.

ELIGIBILITY:
Exclusion Criteria:

* Experience in clinical work with patients
* Prior tonsillectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University first year medical students without any clinical or anatomical experience.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Sufficient intraclass correlation coefficient | At enrollment (day 1)
  The investigators hypothesize that both participants and a trained medical student will be able to assess tonsil size-categorizing them as small, medium, or large, as well as grading them on a 0-4 scale-with sufficient agreement compared to professional evaluation, defined as an intraclass correlation coefficient (ICC) of at least 0.60.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided